CLINICAL TRIAL: NCT07300059
Title: Short-Term Glycemic Effects of Two Concentrations of Liquid Metformin Versus Standard Metformin Tablets in Healthy Adults
Brief Title: Short-Term Glycemic Effects of Liquid Metformin vs Standard Tablets
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASP-020-Met
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Liquid Metformin 100 mg/mL; Drug: Liquid Metformin 250 mg/mL; Drug: Standard Metformin Immediate-Release Tablet

INTERVENTIONS:
Drug: Liquid Metformin 100 mg/mL — A single oral dose of a liquid metformin formulation at a concentration of 100 mg/mL will be administered under fasting conditions in one period of the crossover to assess short-term glycemic effects and safety.
Drug: Liquid Metformin 250 mg/mL — A single oral dose of a liquid metformin formulation at a concentration of 250 mg/mL will be administered under fasting conditions in one period of the crossover to assess short-term glycemic effects and safety.
Drug: Standard Metformin Immediate-Release Tablet — A single oral dose of standard metformin immediate-release tablet(s) will be administered under fasting conditions in one period of the crossover to assess short-term glycemic effects and safety.

SUMMARY:
This is an open-label, randomized study evaluating the short-term glycemic effects of two concentrations of liquid metformin formulations (100 mg/mL and 250 mg/mL) compared with standard immediate-release metformin tablets in healthy adult subjects. Participants will receive single or short-term doses of study treatments in a randomized sequence. Blood glucose measurements and other glycemic indicators will be collected to assess short-term pharmacodynamic effects. Safety and tolerability will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

- Male or female adults 18 to 55 years of age, inclusive.

Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

Medically healthy based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations, in the opinion of the investigator.

Fasting blood glucose within the normal reference range at screening.

Non-smoker or light smoker (10 cigarettes per day or fewer, or equivalent) willing to abstain during each study confinement period.

Able to understand and provide written informed consent before participation.

Willing and able to comply with all study procedures, including fasting requirements, glycemic assessments, and timed blood draws.

Females of childbearing potential must use acceptable contraception as determined by the investigator.

Exclusion Criteria:

* Known hypersensitivity or contraindication to metformin or any excipients in the study formulations.

History or presence of any clinically significant cardiovascular, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or psychiatric condition that, in the investigator's judgment, could interfere with study participation or data interpretation.

Fasting blood glucose outside the normal reference range at screening, or any history of hypoglycemia or glucose regulation disorders.

Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m² or any clinically significant abnormal clinical laboratory results.

History of lactic acidosis.

Use of prescription medications, over-the-counter medications, vitamins, herbal supplements, or dietary supplements within 14 days before first study dosing, unless approved by the investigator.

Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Positive urine drug screen or positive alcohol breath test at screening or admission.

Participation in another clinical study or receipt of an investigational product within 30 days or 5 half-lives (whichever is longer) before the first study dose.

Donation of ≥450 mL of blood, or significant blood loss, within 8 weeks before the first study dose.

Pregnant or breastfeeding females.

Women of childbearing potential not using acceptable contraception.

Any condition that, in the opinion of the investigator, would make the participant unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Blood Glucose-Time Curve from 0 to 4 Hours Postdose (Glucose AUC₀-₄h) | 0 to 4 hours after each study dose in each treatment period

IPD SHARING:
Plan to Share IPD: No